CLINICAL TRIAL: NCT02393612
Title: A Multicenter, Randomized, Double-Blind, Active-Controlled, Parallel Group, Phase III Clinical Trial to Evaluate in Efficacy and Safety of DP-R202 and Anplag Tab in Patients With Artery Occlusive Disease
Brief Title: Clinical Trial to Evaluate Efficacy and Safety of DP-R202 and Anplag in Patients With Artery Occlusive Disease
Acronym: DAVICI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alvogen Korea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DP-CTR202-III-04
Record Dates: First submitted 2015-03-12; First posted 2015-03-19 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2015-03

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DP-R202 (Experimental): Patients administrate DP-R202 (Sarpogrelate 300mg) once a day for 12 weeks
  Interventions: Drug: DP-R202; Drug: Anplag tab
- Anplag tab (Active Comparator): Patients administrate Anplag tab (Sarpogrelate 100mg) 3 times a day for 12 weeks
  Interventions: Drug: DP-R202; Drug: Anplag tab

INTERVENTIONS:
Drug: DP-R202 — Sarpogrelate HCl SR 300mg is administrated to patients with PAD for 12 weeks
  Other Names: Sarpogrelate HCl SR 300mg
Drug: Anplag tab — Anplag tab 100mg is administrated to patients with PAD for 12 weeks

SUMMARY:
Sarpogrelate hydrochloride, a selective 5-HT2A antagonist, has been widely used as an anti-platelet agent for the treatment of PAD. DP-R202 is a new Sarpogrelate hydrochloride product improved patient's convenience and disadvantage of dosage regimen of previous drug. The aim of this study was to compare the efficacy and safety of DP-R202 and Anplag® Tab in patients with PAD

DETAILED DESCRIPTION:
1. Design This clinical trial is 12 weeks, multicenter, randomized, double-blind, parallel group, phase 3 study which registered patients in total 25 institutions appointed as national clinical trial institution, it was conducted by receiving IRB(institutional review board) approval from each institutions.

   Target patients were aged over 20 years old male or female lower limb peripheral artery occlusion patients with fontaine stage II/III, who has lower limb pain or symptoms like leg stretching or numbing, lower limb pain degree is over 40 mm evaluated by VAS at screening, and ABI (ankle-brachial index) ≤0.9 or stenosis rate over >50%, diagnosed with PAD and voluntarily agreed to participate in clinical study and signed study consent form. In addition, exclusion criteria were patients who received peripheral related surgery within 1 month of clinical study participation, Fontaine stage 4, NYHA class 3-4, uncontrollable hypertension patients (systolic BP ≥ 180 mmHg, diastolic BP ≥ 110 mmHg), patients with history of cerebrovascular disease(cerebral infarction, cerebral hemorrhage and etc.) within 6 months prior to clinical trial participation, patients with uncontrollable diabetes (HbA1c ≥ 9%), and patients with renal insufficiency (creatinine > 3.0 mg/dL). Study subjects who met subjects criteria and recruited were total 151 subjects (study group: 75 subjects, comparator group: 76), and among these, 16 subjects (study group: 7 subjects, comparator group: 9 subjects) were dropouts therefore, total study subjects who completed study was 135 subjects (study group: 68 subjects, comparator group: 67 subjects). Dropout reasons were 'clinical trial plan violation' for 3 subjects (comparator group: 3 subjects), ' consent withdrawal' for 8 subjects( study group: 5 subjects, comparator group: 3 subjects), ' fail to follow up' for 1 subject (comparator group: 1 subject), 'adverse event' for 3 subjects ( study group: 1 subject, comparator group: 2 subjects), ' other reasons' for 1 subjects ( study group) and there was no dropout due to 'lack of efficacy'. Selected subjects were stratified by 1:1 ratio and randomly assigned to investigational product or comparator by Fontaine Stage II or Fontaine Stage III using block randomization method and double-blind was applied to both investigator and study subjects.
2. Administration Method Investigational product was DP-R202 (sarpogrelate hydrochloride 300 mg: DreamPharma, Inc.), and comparator was Anplag® Tab (sarpogrelate hydrochloride 100 mg: Yuhan Corp.). Administration period to subjects was 12 weeks, study group took investigational product, DP-R202 1 tab once(morning) and took placebo, Anplag® Tab 1 tab/once, 3 times/day, and comparator group took investigational product, Anplag® Tab 1 tab/once, 3 times/day and took DP-R202, placebo 1 tab once(morning).

   Administration dosage of test drug was conducted as fixed dosage and dosage fluctuation based on subject's condition was not performed.
3. Efficacy and Safety Assessment Parameter Subjects visited at 4, 8, and 12 weeks including baseline visit (visit 2) at 4 weeks interval (total 4 times) and took efficacy and quality of life assessment.

Variation in lower limb pain (VAS) comparing baseline with 12 weeks point as a primary efficacy Assessment parameter, variation in lower limb pain (VAS) and coldness 5-point scale comparing baseline with 4, 8 weeks, ankle brachial pressure index (ABI), ankle systolic pressure (ASP), quality of life assessment index(SF-36), Maximum Walking Distance (MWD), Pain Free Walking Distance (PFWD), and investigator's general assessment(VAS) at 4, 8, and 12 weeks as secondary efficacy assessment parameters, efficacy was measured. Pain and coldness test was measured using pain and coldness felt by subject 24 hours prior to the visit, MWD and PFWD was measured only on subjects who was determined to be possible to measure, and asked to record daily degree of lower limb pain every day from baseline till the end of clinical trial only with subject who can record it. Also, adverse even, laboratory test, vital sign, weight measurement were conducted for efficacy assessment. Physical test and vital sign were conducted at screening visit, administration begins, 4, 8, and 12 weeks after administration and urine pregnancy test and laboratory test were conducted at screening visits and 12 weeks after administration. ECG test was conducted at screening visit, 4, 8, and 12 weeks after administration. Laboratory test criteria were hematological test, blood chemical test, blood coagulation test and urine test.

ELIGIBILITY:
Inclusion Criteria:

* Lower limb pain degree is over 40 mm evaluated by VAS at screening
* ABI (ankle-brachial index) ≤0.9

Exclusion Criteria:

* Patients with peripheral related surgery within 1 month of clinical study participation
* Fontaine stage 4, NYHA class 3-4

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2012-10; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Variation in lower limb pain (VAS) | 12 weeks

IPD SHARING:
Plan to Share IPD: No